CLINICAL TRIAL: NCT00704197
Title: Study of Sex Differences in Characteristics of Adiposity and Metabolism
Brief Title: "ISIS" Study of Sex Differences in Characteristics of Adiposity and Metabolism
Acronym: ISIS
Status: Terminated | Type: Observational
Why Stopped: Study has not been updated since 2016 and PI (Steven R Smith, M.D.) left PBRC. Angela 09/13/2022
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: University of Maryland (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: PBRC 27010
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, urine, adipose tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to characterize differences in the structure and function of the body fat from two different parts of the body in young, healthy men and women. We will also compare how differences in metabolism relate to characteristics of body fat and its functions.

DETAILED DESCRIPTION:
Following screening, the study comprises of a total of 3 clinic visits (2 outpatient visits, and 1 overnight stay) completed during a 2 week period. For the outpatient visits, body composition (by DEXA), visceral fat (by CT), ectopic fat (by MRS and CT) and aerobic fitness (by VO2max test) will be measured. Women will also have ovarian parameters (follicle size and number) measured during the MR scans. Following an overnight stay in the inpatient unit, insulin sensitivity (by euglycemic hyperinsulinemic clamp), interstitial lipolysis (by microdialysis), whole body lipolysis and glycolysis (by stable isotopes), abdominal adipose tissue oxygen content (Hunt and Direct Methods) will be measured and a subcutaneous fat biopsy of the abdominal and gluteo-femoral tissue will be collected. Women will complete all testing in the follicular phase of the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic men and women ages 40 to 60, inclusive and healthy men and women ages 20 to 35, inclusive.
* Body mass index (a ratio of height to weight) less than 25 kg/m2 (lean group) or 27 to 35 kg/m2 (overweight/obese group).
* Not involved in regular physical activity (more than 3 times per week).
* Women must have regular menstrual cycles (1 menstrual bleeding each month).

Exclusion Criteria:

* For men in the overweight/obese group, you have a waist circumference less than 102cm (40 inches).
* You smoke.
* You have liver, kidney, thyroid or heart diseases, or cancer.
* You are claustrophobic.
* You have metal objects in your body such as implanted rods or surgical clips.
* If you are not diabetic and you are taking steroids, protease inhibitors, statins, antihypertensives or medications known to alter glucose or lipid metabolism.
* If you are diabetic and you are taking steroids, protease inhibitors, or injectable antihyperglycemic medications (oral diabetic meds are allowed.)
* If you are a woman, you are pregnant or breast feeding or trying to become pregnant (women who become pregnant throughout the study will be excluded).
* If you are a woman, you are using hormonal contraceptives or have anovulation, androgen excess or irregular menstrual cycles (less than 1 cycle per month).
* You have previously had a BMI >35 kg/m2.
* You are not able to eat the foods provided by PBRC.
* If your weight has not been stable.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of Baton Rouge
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2007-08; Primary Completion 2013-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To assess sex differences in adipose tissue gene expression in different fat depots | baseline

SECONDARY OUTCOMES:
To assess sex differences in other characteristics of adipose tissue structure and function in different fat depots across sex including: preadipocyte kinetics; lipolysis and lipogenesis; macrophage content; and tissue oxygenation | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Nunez Lopez YO, Garufi G, Pasarica M, Seyhan AA. Elevated and Correlated Expressions of miR-24, miR-30d, miR-146a, and SFRP-4 in Human Abdominal Adipose Tissue Play a Role in Adiposity and Insulin Resistance. Int J Endocrinol. 2018 Mar 12;2018:7351902. doi: 10.1155/2018/7351902. eCollection 2018. PMID 29721017
- [Derived] Divoux A, Xie H, Li JL, Karastergiou K, Perera RJ, Chang RJ, Fried SK, Smith SR. MicroRNA-196 Regulates HOX Gene Expression in Human Gluteal Adipose Tissue. Obesity (Silver Spring). 2017 Aug;25(8):1375-1383. doi: 10.1002/oby.21896. Epub 2017 Jun 25. PMID 28649807
- [Derived] Pasarica M, Rood J, Ravussin E, Schwarz JM, Smith SR, Redman LM. Reduced oxygenation in human obese adipose tissue is associated with impaired insulin suppression of lipolysis. J Clin Endocrinol Metab. 2010 Aug;95(8):4052-5. doi: 10.1210/jc.2009-2377. Epub 2010 May 13. PMID 20466783